CLINICAL TRIAL: NCT01214200
Title: High Intensity Non-Invasive Positive Pressure Ventilation (HINPPV) for Stable Hypercapnic Chronic Obstructive Pulmonary Disease (COPD) Patients
Brief Title: High Intensity Non-Invasive Positive Pressure Ventilation (HINPPV)
Acronym: HINPPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRC-0927-HINPPV-MS
Record Dates: First submitted 2010-06-29; First posted 2010-10-04 (Estimated); Results first posted 2019-01-02 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- High Intensity Non Invasive Pos.Pressure (Experimental): The High Intensity Non-invasive Pos.Pressure trial is a single arm interventional study. Hypercapnic COPD participants that meet eligibility criteria will receive high intensity non-invasive positive pressure ventilation (HINPPV) for 90 days. Participants will receive HINPPV via bilevel positive airway pressure (BiPAP Synchrony) if they require an inspiratory positive airway pressure (IPAP) less than or equal to 30 cmH2O (centimeters of water); or the Trilogy ventilator if they require an IPAP greater than 30 cmH2O.
  Interventions: Device: Bilevel positive airway pressure (BiPAP)

INTERVENTIONS:
Device: Bilevel positive airway pressure (BiPAP) — This is a single arm interventional study. Hypercapnic COPD participants that meet eligibility criteria will receive high intensity non-invasive positive pressure ventilation(HINPPV). Participants will receive HINPPV via bilevel positive airway pressure (BiPAP) via a Synchrony ventilator if they require an inspiratory positive airway pressure (IPAP) less than or equal to 30 cmH2O; or the Trilogy ventilator if they require an IPAP greater than 30 cmH2O.
  Other Names: Synchrony BiPAP ventilator and Trilogy Ventilator

SUMMARY:
The purpose of this pilot study is to evaluate the effect of high intensity non-invasive positive pressure ventilation (HINPPV) for stable, hypercapnic COPD patients. The investigators believe that HINPPV, used at least 6 hours nocturnally over three months, will benefit the stable hypercapnic COPD patient through a reduction in the daytime partial pressure of carbon dioxide in arterial blood (PaCO2) levels.

DETAILED DESCRIPTION:
The High Intensity Non-invasive Positive Pressure trial is a single arm interventional study. The purpose of this study is to evaluate the effect of High Intensity Non-invasive ventilation (HINPPV) in stable Chronic Obstructive Pulmonary patients with chronically elevated carbon dioxide levels. Participants will undergo various testing ( arterial blood gas (ABG), Pulmonary Function Test (PFTs), Polysomnography (PSGs), 6 minute walk tests)over a 3 month period to determine if this type of therapy will improve daytime carbon dioxide levels. The participants will also complete quality of life questionnaires to help ascertain improvements in their daily living activities.

ELIGIBILITY:
Inclusion Criteria

1. Patient diagnosed with chronic obstructive pulmonary disease (COPD)
2. Age < or = to 80 years
3. Forced expiratory volume in one second (FEV1) < 50% of predicted value
4. FEV1/Forced vital capacity (FVC) < 70% of predicted value
5. Total lung capacity (TLC) > 90% predicted by plethysmography
6. Body Mass Index (BMI) < 35
7. Patient has provided written informed consent using a form that has been approved by the Internal Review Board (IRB)
8. Daytime PaCO2 ≥ 52 mm Hg, at rest on room air (Denver > 48 mm Hg) with one of the following symptoms of hypercapnia:

   * Fatigue
   * Sleepiness
   * Headaches
9. Post hospital discharge at least one month prior to screening visit
10. Participant is willing and able to complete all required assessments and procedures
11. Participant has no child bearing potential OR a negative pregnancy test in a woman of childbearing potential

Exclusion Criteria

1. FEV1 < 15% of predicted value
2. Diagnosis of obstructive sleep apnea (OSA) [Apnea hypopnea index (AHI) > 15 per hour]
3. Current Non-invasive Positive Pressure Ventilation (NIPPV), Positive Airway Pressure (PAP) or Non-invasive Ventilation (NIV) users
4. Signs / symptoms of acute exacerbation within the previous month: two of the following criteria:

   * Increasing cough
   * Purulent sputum
   * Current use of antibiotics
   * pH < 7.35
5. Any major non COPD disease or condition that interferes with completion of initial or follow-up assessments, such as uncontrolled malignancy, end-stage heart disease, liver or renal insufficiency (that requires current evaluation for liver or renal transplantation or dialysis), amyotrophic lateral sclerosis, or severe stroke, or other as deemed appropriate by investigator as determined by review of medical history and / or patient reported medical history
6. History of pneumothorax
7. Anatomical facial abnormalities precluding placement of a nasal or facial mask
8. Diffuse parenchymal lung disease other than emphysema
9. Inability to maintain Oxygen (O2) saturation >90% on 5L/min ( five liters) nasal O2 at rest
10. Sustained need for >10 mg prednisone daily or equivalent dose of other systemic corticosteroid
11. Pregnancy
12. Excessive alcohol intake (≥ 6oz hard liquor daily), or illicit drug use
13. Daily use of narcotics (greater than 30 mg morphine equivalent)
14. Patient is currently enrolled in another interventional clinical trial

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Criner, MD, Principal Investigator — Temple Medical Center
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- High Intensity Non Invasive Pos.Pressure: The High Intensity Non-invasive Positive Pressure (HINPPV) trial is a single arm interventional study. Hypercapnic Chronic Obstructive Pulmonary Diseased (COPD) participants that meet eligibility criteria will receive HINPPV for 90 days. Participants will receive HINPPV via bilevel positive airway pressure (BiPAP Synchrony) if they require an inspiratory positive airway pressure (IPAP) less than or equal to 30 cmH2O (centimeters of water); or the Trilogy ventilator if they require an IPAP greater than 30 cmH2O.
Period: Overall Study
Arm/Group | High Intensity Non Invasive Pos.Pressure
Started | 20
Completed | 9
Not Completed | 11
Not completed — Did not meet inclusion/exclusion | 9
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Demographics were only evaluated on those that consented and completed the trial.
Groups:
- High Intensity Non Invasive Pos.Pressure: The High Intensity Non-invasive Positive Pressure (HINPPV) trial is a single arm interventional study. Hypercapnic COPD participants that meet eligibility criteria will receive HINPPV) for 90 days. Participants will receive HINPPV via bilevel positive airway pressure (BiPAP Synchrony) if they require an inspiratory positive airway pressure (IPAP) less than or equal to 30 cmH2O; or the Trilogy ventilator if they require an IPAP greater than 30 cmH2O.
Arm/Group | High Intensity Non Invasive Pos.Pressure
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9
Forced Expiratory Volume 1 sec (FEV1s) [Mean (Standard Deviation); unit: percent of predicted] | 26 (6.73)
BMI [Mean (Inter-Quartile Range); unit: kg/m^2] | 26.6 [25.5 to 32.5]
Cigarette Usage [Median (Inter-Quartile Range); unit: packs per year] | 55 [45 to 90]

OUTCOME MEASURES:

1. Primary Outcome: Daytime Partial Pressure of Carbon Dioxide in Arterial Blood (PaCO2)
Description: Daytime PaCO2 levels assessed after using high intensity non-invasive positive pressure ventilation (HINPPV) are compared to the participants' baseline daytime PaCO2 levels.
Time Frame: Before and after 3 months of therapy
Measure: Mean (Inter-Quartile Range); unit: mmHg
Arm/Group | High Intensity Non Invasive Pos.Pressure
Number analyzed (Participants) | 9
mmHg
  Baseline | 53 [52.9 to 60.5]
  3 months | 50 [47.5 to 54.5]
Statistical Analysis 1: Comparison: High Intensity Non Invasive Pos.Pressure; Test type: Other — For the analysis of differences between pre and post treatment a student's t-test was used and was checked with the Wilcoxon signed rank test. A p<0.05 was considered statistically significant; p = 0.01, Wilcoxon Signed Ranks Test

2. Secondary Outcome: Health Status
Description: Health status was assessed by completing different surveys at baseline and after 3 months of therapy. The Calgary Sleep Apnea Quality of Life was administered at baseline and 3 months. It is a 35-item, interview-administered scale, the SAQLI evaluates four domains of quality of life associated with sleep apnea: daily functioning, social interactions, emotional functioning, and symptoms. The SAQLI use a 7-point Likert scale ranging from 1 (maximal impairment) to 7 (no impairment).
Time Frame: Before and after 3 months of therapy
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | High Intensity Non Invasive Pos.Pressure
Number analyzed (Participants) | 9
units on a scale
  Baseline | 4.34 [3.44 to 5.6]
  3 months | 4.78 [4.64 to 5.6]

3. Secondary Outcome: Maximal Inspiratory Pressure
Description: The Maximal inspiratory pressure (MIP) is the maximum negative pressure that can be generated from one inspiratory effort starting from functional residual capacity (FRC) or residual volume (RV). This was assessed at baseline and after 3 months of therapy.
Time Frame: Before and after 3 months of therapy
Measure: Mean (Inter-Quartile Range); unit: kPa
Arm/Group | High Intensity Non Invasive Pos.Pressure
Number analyzed (Participants) | 9
kPa
  Baseline | 7.04 [3.67 to 7.97]
  3 months | 6.85 [3.9 to 8.3]

4. Secondary Outcome: Exercise Capacity
Description: Exercise capacity will be measured by comparing the 6 minute walk test as measured in meters from baseline to 3 months
Time Frame: Before and after 3 months of therapy
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | High Intensity Non Invasive Pos.Pressure
Number analyzed (Participants) | 9
meters
  Baseline | 211 (54)
  3 months | 236 (80)

5. Secondary Outcome: Dyspnea at Rest and With Exertion
Description: The modifed Borg scale was used to measure dyspnea. The Dyspnea Borg scale measures patients perceived level of dyspnea. The scale ranges from 0 to 10, 0- nothing at all and 10 is maximal.
Time Frame: Before and after 3 months of therapy
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- At Rest: All participants competed the modifed Borg scale at rest, prior to exercise.
- After Exertion: All participants completed the modified Borg scale after exertion (6 minute walk test).
Arm/Group | At Rest | After Exertion
Number analyzed (Participants) | 9 | 9
units on a scale
  Baseline | 0.7 (1.3) | 6.9 (1.7)
  3 months | 0.6 (1.1) | 4.6 (1.7)

6. Secondary Outcome: Sleepiness
Description: Sleepiness will be evaluated by measuring the the baseline and 3 month Epworth Sleepiness Scale. The Epworth Sleepiness Scale is an 8 question survey regarding daytime sleepiness. The higher the score the higher the chance of dozing during the day. Each question is rated on a 0 to 3 scale of chance of dozing or sleeping. 0 would be no chance, 3 would be the highest chance.
Time Frame: Before and after 3 months of therapy
Population: Only 5 participants completed the overnight polysomnography (PSG) for this trial.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Intensity Non Invasive Pos.Pressure
Number analyzed (Participants) | 5
units on a scale
  Baseline | 9.3 (2.6)
  3 months | 7.2 (3.3)

7. Secondary Outcome: Duration of Sleep
Description: Duration of sleep will be measured using total sleep time. Total sleep time is the overall number of minutes of sleep, this will be compared from baseline to 3 months.
Time Frame: Before and after 3 months of therapy
Population: Only 5 participants completed the overnight PSG for this trial.
Measure: Mean (Standard Deviation); unit: minutes per night
Arm/Group | High Intensity Non Invasive Pos.Pressure
Number analyzed (Participants) | 5
minutes per night
  Baseline | 329 (62.5)
  3 months | 337 (34)

8. Secondary Outcome: Efficiency of Sleep
Description: Sleep efficiency will be measured by taking the total sleep time by the total time in bed. This is measured as a percentage and compared from baseline to 3 months
Time Frame: Before and after 3 months of therapy
Population: Only 5 participants completed the overnight PSG for this trial.
Measure: Mean (Standard Deviation); unit: percentage of efficiency
Arm/Group | High Intensity Non Invasive Pos.Pressure
Number analyzed (Participants) | 5
percentage of efficiency
  Baseline | 80.6 (12.7)
  3 months | 83.6 (6.7)

ADVERSE EVENTS:
Arm/Group | High Intensity Non Invasive Pos.Pressure
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 4/9
Other Adverse Events (participants affected / at risk) | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Intensity Non Invasive Pos.Pressure (N=9)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No